CLINICAL TRIAL: NCT06578221
Title: The Effects of Kegel Pelvic Floor Muscle Exercises on Urinary Retention and Comfort Level of Patients After Lumbar Disc Herniation Surgery: A Randomised Controlled Trial
Brief Title: The Effects of Kegel Pelvic Floor Muscle Exercises on Urinary Retention and Comfort Levels
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Büşra Demirci, Principal İnvestigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15151515
Record Dates: First submitted 2024-08-14; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Nurses; Comfort; Surgery
Keywords: Nurses; İntervertebral Disc; Comfort; Patient Urinary Retention; Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kegel Pelvic Floor Muscle Exercise Group (Experimental): Kegel exercises will be performed by the researcher within the first 8 hours after being taken to the clinic room to perform the Kegel pelvic floor muscle exercises while in the supine position. Urinary retention and comfort level of patients will be evaluated after surgery.
  Interventions: Other: Kegel Pelvic Floor Muscle Exercise Group
- Control Group (No Intervention): Urinary retention and comfort level of patients will be evaluated after surgery.

INTERVENTIONS:
Other: Kegel Pelvic Floor Muscle Exercise Group — After the surgery, the patients will be taken to the clinic room in a supine position and the researcher will perform the Kegel pelvic floor muscle exercises three times at the 1st, 4th and 7th hours within the first 8 hours after the patients are taken to the clinic room.
  Arms: Kegel Pelvic Floor Muscle Exercise Group

SUMMARY:
This study was planned as a randomized controlled trial to investigate the effects of Kegel pelvic floor muscle exercises on urinary retention and comfort levels of patients after lumbar disc herniation surgery.

DETAILED DESCRIPTION:
Postoperative urinary retention is the inability to urinate despite having a full bladder after surgery. It is a relatively common complication of both outpatient and inpatient procedures. Most cases are transient and are managed by temporarily emptying the bladder with bladder catheterization.

Studies in the literature report that transient postoperative urinary retention is common after cervical and lumbar spine surgery procedures. This situation is of great importance in terms of healthcare services, as it can increase both the length of hospital stay and the cost.

Kegel pelvic floor muscle exercises involve the repeated contraction and relaxation of the muscles that form part of the pelvic floor. With these exercises, pelvic floor blood circulation can be increased, pelvic floor muscle tension can be increased, and the contraction of the relaxed bladder can be stimulated indirectly by repeated contraction and relaxation of the pelvic floor muscles, and urine output can be achieved. Therefore, we think that these exercises, which are safe, cost-effective exercises that can be easily applied by healthcare personnel, and patient comfort among nursing practices to improve perioperative results and functional status, will have an effect in preventing urinary retention.

There are no experimental studies in the literature evaluating the effect of Kegel exercises applied after lumbar disc herniation surgery on urinary retention. Therefore, this study was planned to be conducted in patients who will undergo lumbar disc herniation surgery.

This study was planned as a single-center prospective randomized controlled experimental study. After obtaining verbal and written consent from the patients before surgery, the study will be conducted with various data collection forms.

These forms; Patient Information Form, Postoperative Data Collection Form, Numeric Rating Scale (NRS) to determine the pain level of the patients and Visual Analog Scale (VAS) to evaluate the comfort level. Patients will be randomized. Group I will be the Kegel pelvic floor muscle exercise group (n=29), Group II will be the control group (n=29). It is planned to measure the urinary retention and comfort levels of both groups in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study
* Over 18 years of age
* No communication barrier
* Having undergone lumbar disc herniation surgery under general anesthesia
* Being immobile for the first 8 hours postoperatively
* Not having a urinary catheter inserted during the intraoperative period

Exclusion Criteria:

* Refusal to participate in the study
* Previous urinary disorders/symptoms (such as Benign Prostatic Hyperplasia)
* Spinal trauma, preoperative neurological disorder
* Patients with preoperative catheterization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Having had surgery for lumbar disc herniation
Enrollment: 58 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Effect of Kegel pelvic floor muscle exercises on urinary retention of patients after lumbar disc herniation surgery. | After completing Kegel pelvic floor muscle exercises in the first 8 hours after surgery.
  Kegel pelvic floor muscle exercises will affect the urinary retention of patients after lumbar disc herniation surgery. This situation will be evaluated with the Postoperative Data Collection Form. The Postoperative Data Collection form, which was created by the researchers as a result of a literature review, includes a total of 10 questions including postoperative pain, vital signs, and postoperative (postoperative first 8 hours) urinary retention signs and symptoms (pressure in the lower abdomen, pain in the lower abdomen, feeling of restlessness, desire to urinate within 8 hours?).

SECONDARY OUTCOMES:
Effect of Kegel pelvic floor muscle exercises on comfort level after lumbar disc herniation surgery | After completing Kegel pelvic floor muscle exercises in the first 8 hours after surgery.
  Kegel pelvic floor muscle exercises will affect comfort level of patients after lumbar disc herniation surgery. The comfort level of the patients will be evaluated with VAS. VAS is used to convert some unmeasurable values into numerical values. VAS is a horizontal line with a length of 10 cm. According to VAS, 0 is the lowest level and 10 is the highest level. Patients will be asked to mark these levels on the 10 cm line.

CONTACTS AND LOCATIONS:
Locations (1):
- Büşra Demirci, Ankara, University of Health Sciences, Turkey (Türkiye)

REFERENCES:
- [Background] Pomajzl AJ, Siref LE. Postoperative Urinary Retention. 2023 Jul 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK549844/ PMID 31751034
- [Background] Wang R, Tunitsky-Bitton E. Short-term catheter management options for urinary retention following pelvic surgery: a cost analysis. Am J Obstet Gynecol. 2022 Jan;226(1):102.e1-102.e9. doi: 10.1016/j.ajog.2021.07.025. Epub 2021 Aug 5. PMID 34363780
- [Background] Altschul D, Kobets A, Nakhla J, Jada A, Nasser R, Kinon MD, Yassari R, Houten J. Postoperative urinary retention in patients undergoing elective spinal surgery. J Neurosurg Spine. 2017 Feb;26(2):229-234. doi: 10.3171/2016.8.SPINE151371. Epub 2016 Oct 21. PMID 27767680
- [Background] Aiyer SN, Kumar A, Shetty AP, Kanna RM, Rajasekaran S. Factors Influencing Postoperative Urinary Retention Following Elective Posterior Lumbar Spine Surgery: A Prospective Study. Asian Spine J. 2018 Dec;12(6):1100-1105. doi: 10.31616/asj.2018.12.6.1100. Epub 2018 Oct 16. PMID 30322244
- [Background] Boulis NM, Mian FS, Rodriguez D, Cho E, Hoff JT. Urinary retention following routine neurosurgical spine procedures. Surg Neurol. 2001 Jan;55(1):23-7; discussion 27-8. doi: 10.1016/s0090-3019(01)00331-7. PMID 11248301
- [Background] Boonstra AM, Schiphorst Preuper HR, Reneman MF, Posthumus JB, Stewart RE. Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. Int J Rehabil Res. 2008 Jun;31(2):165-9. doi: 10.1097/MRR.0b013e3282fc0f93. PMID 18467932